CLINICAL TRIAL: NCT01432639
Title: Effects of Exercise Training on Endothelial Function, Inflammation, Arterial Stiffness and Autonomic Function in Coronary Artery Disease Patients
Brief Title: Effects of Exercise Training on Endothelial Function, Inflammation, Arterial Stiffness and Autonomic Function in CAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Centro Hospitalar de Vila Nova de Gaia/Espinho (Other); Research Center in Physical Activity, Health and Leisure, Portugal (Unknown)
Responsible Party: Principal Investigator, Jose Manuel Fernandes Oliveira, Professor, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTDC/DES/113753/2009
Record Dates: First submitted 2011-09-07; First posted 2011-09-13 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Coronary Artery Disease
Keywords: Myocardial infarction; Autonomic function; Arterial Stiffness; Endothelial function; Inflammation; Rehabilitation program; Exercise
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Inflammation; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): Patients undergoing the exercise-based cardiac rehabilitation program (intervention)
  Interventions: Other: Exercise-based cardiac rehabilitation program
- Control group (No Intervention): Usual medical care

INTERVENTIONS:
Other: Exercise-based cardiac rehabilitation program — The intervention consists of usual medical care (i.e., medicine prescription and counseling of lifestyle modifications) and an supervised outpatient aerobic exercise training, which will be performed 3 days per week for 8 weeks. Each exercise session include 10 min of warm up, 35 min of aerobic exercise (i.e., cycloergometer or treadmill) and 10 min of cool down. The exercise intensity will be calculated as 65- 75% of maximal heart rate achieved in the treadmill exercise testing. Individualized exercise prescription will be periodically adjusted. A perceived exertion scale will be used as an adjunctive intensity modulator. In addition, each patient will be encouraged to daily exercise outside the formal exercise program.
  Other Names: Cardiac rehabilitation program
  Arms: Experimental group

SUMMARY:
The main purposes of this study is to analyze, in a randomized controlled trial, the effects of an exercise-based cardiac rehabilitation program (i) on biomarkers of endothelial function, (ii) on biomarkers of inflammation, (iii) on autonomic function, and (iv) on arterial stiffness in coronary artery disease patients (CAD). Additionally, the investigators aim to analyze the (v) contribution of age and the changes in traditional risk factors to the modification of the endothelial dysfunction and inflammation, and (vi) the contribution of the changes in inflammatory and endothelial function biomarkers to the modification of autonomic function and arterial stiffness.

The investigators hypothesize that exercise training will improve the autonomic function, arterial stiffness and mitigate the endothelial dysfunction and inflammation in CAD patients even in the absence of significant changes in traditional risk factors. Thus, the investigators expect with the present study to promote, develop and expand the knowledge in this field by assessing the impact of exercise on a pool of markers that provide a wide picture of the pathophysiological processes underlying CAD.

ELIGIBILITY:
Inclusion Criteria:

* acute myocardial infarction

Exclusion Criteria:

* ventricular tachyarrhythmia
* uncontrolled hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure >100 mmHg)
* significant valvular disease
* unstable angina pectoris
* reduced left ventricular function (ejection fraction < 45%)
* abnormal hemodynamic response
* myocardial ischemia and/or severe ventricular arrhythmias during baseline exercise testing
* uncontrolled metabolic disease (e.g. uncontrolled diabetes or thyroid disease)
* presence of pulmonary and renal co-morbidities
* peripheral artery disease and/or orthopedic limitations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Autonomic Function | Change from Baseline in Autonomic Function at 8 weeks of Cardiac Rehabilitation Program
  Autonomic function will be assessed by resting heart rate variability, heart rate recovery after maximal exercise and circulating levels of norepinephrine and epinephrine.

SECONDARY OUTCOMES:
Arterial Stiffness | Change from Baseline in Arterial Stiffness at 8 weeks of Cardiac Rehabilitation Program
  Arterial Stiffness will be assessed by carotid-femoral pulse wave velocity and the aortic augmentation index.
Endothelial Function | Change from Baseline in Endothelial Function at 8 weeks of Cardiac Rehabilitation Program
  Using commercially available assay kits (R&D Systems, Minneapolis, MN, USA), the serum levels of sICAM-1 and sVCAM-1 will be measured in serum by an enzyme-linked immunosorbent assay (ELISA) according to the manufacturer's instructions and read at 450 nm using a microplate reader (Labsystems iEMS MF controlled by Ascent software v. 2.4, Dynex Labsystems).
Cardiorespiratory Fitness | Change from Baseline in Cardiorespiratory Fitness at 8 weeks of Cardiac Rehabilitation Program
  Maximal or symptom-limited treadmill exercise testing will be conducted using the modified Bruce protocol.
Inflammatory Biomarkers | Change from Baseline in Inflammatory Biomarkers at 8 weeks of Cardiac Rehabilitation Program
  Using commercially available assay kits (R&D Systems, Minneapolis, MN, USA), the serum levels of CRP, IL-10 and IL-6 will be measured in serum by an enzyme-linked immunosorbent assay (ELISA) according to the manufacturer's instructions and read at 450 nm using a microplate reader (Labsystems iEMS MF controlled by Ascent software v. 2.4, Dynex Labsystems).
Anthropometrics | Change from Baseline in Anthropometrics at 8 weeks of Cardiac Rehabilitation Program
  Height and weight measurements will be assessed using a standard wall-mounted stadiometer and portable digital beam scale (SECA, 708), respectively. Body mass index will be calculated from the ratio of weight (kg) to squared height (m2). Percentage of fat mass will be estimated by bioelectrical impedance analysis (BC-532, Tanita, Tokyo, Japan).
Blood Pressure | Change from Baseline in Blood Pressure at 8 weeks of Cardiac Rehabilitation Program
  Resting systolic and diastolic blood pressure will be measured using a digital automatic blood pressure monitor (Omron Pressmate BP10, Omron Healthcare Co., Ltd, Kyoto, Japan).
Dietary Intake | Change from Baseline in Dietary Intake at 8 weeks of Cardiac Rehabilitation Program
  Dietary intake will be assessed using a 4-day food diary as representative of the usual intake. Patients will be asked to provide detailed information concerning the food and beverages intake for four days (Sunday and 3-week days).
Daily Physical Activity | Change from Baseline in Daily Physical Activity at 8 weeks of Cardiac Rehabilitation Program
  Physical activity will be objectively measured for 7 consecutive days using the ActiGraph accelerometer (model GT1M, Florida, USA).
Biochemical Parameters | Change from Baseline in Biochemical Parameters at 8 weeks of Cardiac Rehabilitation Program
  Fasting plasma glucose, total cholesterol, high-density lipoprotein cholesterol, triglycerides, and HbA1c will be measured by enzymatic methods (912 automatic analyzer, Roche Diagnostic, Basel, Switzerland). Low-density lipoprotein cholesterol will be calculated using the Friedewald equation, except if triglycerides > 400 mg/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Oliveira, PhD, Study Chair — Research Center in Physical Activity, Health and Leisure, Portugal; Fernando Ribeiro, PhD, Study Director — Research Center in Physical Activity, Health and Leisure, Portugal; Nórton L Oliveira, MSc, Principal Investigator — Research Center in Physical Activity, Health and Leisure, Portugal; Madalena Teixeira, MD, Principal Investigator — Centro Hospitalar de Vila Nova de Gaia/Espinho
Locations (1):
- Centro Hospitalar de Vila Nova de Gaia/Espinho, Vila Nova de Gaia, Portugal

REFERENCES:
- [Background] Ribeiro F, Alves AJ, Duarte JA, Oliveira J. Is exercise training an effective therapy targeting endothelial dysfunction and vascular wall inflammation? Int J Cardiol. 2010 Jun 11;141(3):214-21. doi: 10.1016/j.ijcard.2009.09.548. Epub 2009 Nov 6. PMID 19896741
- [Background] Graham LN, Smith PA, Stoker JB, Mackintosh AF, Mary DA. Time course of sympathetic neural hyperactivity after uncomplicated acute myocardial infarction. Circulation. 2002 Aug 13;106(7):793-7. doi: 10.1161/01.cir.0000025610.14665.21. PMID 12176949
- [Background] Laing ST, Gluckman TJ, Weinberg KM, Lahiri MK, Ng J, Goldberger JJ. Autonomic effects of exercise-based cardiac rehabilitation. J Cardiopulm Rehabil Prev. 2011 Mar-Apr;31(2):87-91. doi: 10.1097/HCR.0b013e3181f1fda0. PMID 20861747
- [Background] Sandercock GR, Grocott-Mason R, Brodie DA. Changes in short-term measures of heart rate variability after eight weeks of cardiac rehabilitation. Clin Auton Res. 2007 Feb;17(1):39-45. doi: 10.1007/s10286-007-0392-5. Epub 2007 Feb 6. PMID 17285225
- [Background] Weber T, Auer J, O'rourke MF, Kvas E, Lassnig E, Lamm G, Stark N, Rammer M, Eber B. Increased arterial wave reflections predict severe cardiovascular events in patients undergoing percutaneous coronary interventions. Eur Heart J. 2005 Dec;26(24):2657-63. doi: 10.1093/eurheartj/ehi504. Epub 2005 Sep 23. PMID 16183688
- [Background] Edwards DG, Schofield RS, Magyari PM, Nichols WW, Braith RW. Effect of exercise training on central aortic pressure wave reflection in coronary artery disease. Am J Hypertens. 2004 Jun;17(6):540-3. doi: 10.1016/j.amjhyper.2003.12.001. PMID 15177529
- [Background] Psychari SN, Apostolou TS, Iliodromitis EK, Kourakos P, Liakos G, Kremastinos DT. Inverse relation of C-reactive protein levels to heart rate variability in patients after acute myocardial infarction. Hellenic J Cardiol. 2007 Mar-Apr;48(2):64-71. PMID 17489343
- [Background] Chesterton LJ, Sigrist MK, Bennett T, Taal MW, McIntyre CW. Reduced baroreflex sensitivity is associated with increased vascular calcification and arterial stiffness. Nephrol Dial Transplant. 2005 Jun;20(6):1140-7. doi: 10.1093/ndt/gfh808. Epub 2005 Apr 12. PMID 15827047
- [Derived] Oliveira NL, Ribeiro F, Silva G, Alves AJ, Silva N, Guimaraes JT, Teixeira M, Oliveira J. Effect of exercise-based cardiac rehabilitation on arterial stiffness and inflammatory and endothelial dysfunction biomarkers: a randomized controlled trial of myocardial infarction patients. Atherosclerosis. 2015 Mar;239(1):150-7. doi: 10.1016/j.atherosclerosis.2014.12.057. Epub 2015 Jan 14. PMID 25602857
- [Derived] Oliveira NL, Ribeiro F, Teixeira M, Campos L, Alves AJ, Silva G, Oliveira J. Effect of 8-week exercise-based cardiac rehabilitation on cardiac autonomic function: A randomized controlled trial in myocardial infarction patients. Am Heart J. 2014 May;167(5):753-61.e3. doi: 10.1016/j.ahj.2014.02.001. Epub 2014 Feb 17. PMID 24766987